CLINICAL TRIAL: NCT07162740
Title: Comparative Study of Right Atrial Versus Bi-atrial Cardioneuroablation of Asystolic Reflex Syncope Verified by Implantable Loop Recorder
Brief Title: Implantable Loop Recorder and Cardioneuroblation
Acronym: ILR-CNA
Status: Not yet recruiting | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: ILR-CNA
Record Dates: First submitted 2025-08-01; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Reflex Syncope
Keywords: Syncope; reflex syncope; implantable loop recorder; Vagal ganglia ablation; Cardioneuroablation; Asystole
MeSH Terms: conditions — Syncope, Vasovagal; Syncope; Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Right atrial ablation group
  Interventions: Procedure: Right atrial ablation
- Bi-atrial ablation group
  Interventions: Procedure: Bi-atrial ablation

INTERVENTIONS:
Procedure: Right atrial ablation — Eligible patients receive the implantation of a LuxDx® ILR and are monitored for one month by means of the Latitude Clarity data management system of the device. The usual practice of the centres is unchanged. According to their usual practice, the centre is assigned to right atrial ablation. The patients receive a right atrial procedure accordingly. As per pragmatic design, cross-over are permitted according to investigator judgment. The ablation methods and techniques are left to investigator's decision. They are reported in the CRF.
  Groups: Right atrial ablation group
Procedure: Bi-atrial ablation — Eligible patients receive the implantation of a LuxDx® ILR and are monitored for one month by means of the Latitude Clarity data management system of the device. The usual practice of the centres is unchanged. According to their usual practice, the centre is assigned to bi-atrial ablation. The patients receive a bi-atrial procedure accordingly. As per pragmatic design, cross-over are permitted according to investigator judgment. The ablation methods and techniques are left to investigator's decision. They are reported in the CRF.
  Groups: Bi-atrial ablation group

SUMMARY:
The study aims to determine which method of vagal ganglia ablation is most effective in preventing recurrences of reflex asystole syncope. Currently, some centers perform ablation only in the right atrium, others in both atria (biatrial). There are no comparative studies between the two procedures

DETAILED DESCRIPTION:
Cardioneuroablation (CNA) therapy for reflex asystole syncope is becoming increasingly popular. The best method of CNA is debated, with no studies comparing the syncopal recurrence rates of right atrium ablation versus bi-atrial ablation. Evaluating the clinical efficacy of CNA is challenging due to symptom variability, intermittent presentation, complex pathophysiology, and different treatment options. The difficulty of obtaining precise follow-up data in patients with intermittent symptoms is well known. With ILR, more objective tracking can be achieved.

The aim of the study is to verify the efficacy of CNA on the reduction of the asystole reflex documented by continuous monitoring by ILR in patients undergoing right atrial ablation compared to bi-atrial ablation

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 60 years
* Clinical diagnosis of reflex syncope as per class I criteria of the ESC guidelines
* History of recurrent severe syncopes (≥2 in the last year or ≥3 in the last 2 years), significantly affecting the quality of life, nonresponding to lifestyle measures.
* Documentation by means of prolonged ECG monitoring of an asystolic pause >6 sec or of an asystolic syncope >3 sec and/or an asystolic syncope induced during tilt testing (Vasis 2B form).

Exclusion Criteria:

* Intrinsic sinus dysfunction or atrioventricular node disease.
* Constitutional hypotension and orthostatic intolerance syndromes
* Overt structural heart disease
* Alternative diagnoses of syncope
* Pregnancy or breastfeeding

Ages: 18 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Established asystolic reflex syncope
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Mounthly frequency of asystolic episodes >3 sec | through study completion, an average of 1 year
  Frequency of asystolic episodes >3 sec per month detected through ILR monitoring before and after ablation.
Freedom from ablation-related complications | through study completion, an average of 1 year
  Freedom from ablation-related complications and from pacemaker implantation during the follow-up period;

SECONDARY OUTCOMES:
Burden of syncopal episodes | through study completion, an average of 1 year
  Comparison betwen the mounthly burden of syncopal episodes before and after ablation;
heart rate (HR) and heart rate variability (HRV) | through study completion, an average of 1 year
  Pattern of heart rate (HR) and heart rate variability (HRV) detected by ILR before andafter ablation.
Time to first asystolic and syncope recurrence | through study completion, an average of 1 year
  Tme to first asystolic pause >3 sec e and to first syncope recurrence

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Auxologico Italiano, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes
After 6 months from the publication of the study upon reasonable request

REFERENCES:
- [Result] Kulakowski P, Baran J, Sikorska A, Krynski T, Niedzwiedz M, Soszynska M, Piotrowski R. Cardioneuroablation for reflex asystolic syncope: Mid-term safety, efficacy, and patient's acceptance. Heart Rhythm. 2024 Mar;21(3):282-291. doi: 10.1016/j.hrthm.2023.11.022. Epub 2023 Nov 29. PMID 38036236
- [Result] Calo L, Rebecchi M, De Ruvo E, Giamundo D, Sette A, Tomaino M, Hunteruber M, Bottoni N, Iori M, Donateo P, Maggi R, Del Rosso A, Rafanelli M, Russo V, Strano S, Brignole M. Right atrial cardioneuroablation of asystolic reflex syncope. Heart Rhythm. 2025 Oct;22(10):e951-e958. doi: 10.1016/j.hrthm.2025.05.038. Epub 2025 May 22. PMID 40412604
- [Result] Aksu T, Brignole M, Calo L, Debruyne P, Di Biase L, Deharo JC, Fanciulli A, Fedorowski A, Kulakowski P, Morillo C, Moya A, Piotrowski R, Stec S, Sutton R, van Dijk JG, Wichterle D, Tse HF, Yao Y, Sheldon RS, Vaseghi M, Pachon JC, Scanavacca M, Meyer C, Amin R, Gupta D, Magnano M, Malik V, Schauerte P, Shen WK, Acosta JCZ. Cardioneuroablation for the treatment of reflex syncope and functional bradyarrhythmias: A Scientific Statement of the European Heart Rhythm Association (EHRA) of the ESC, the Heart Rhythm Society (HRS), the Asia Pacific Heart Rhythm Society (APHRS) and the Latin American Heart Rhythm Society (LAHRS). Europace. 2024 Aug 3;26(8):euae206. doi: 10.1093/europace/euae206. PMID 39082698